CLINICAL TRIAL: NCT00772304
Title: Evaluation of the Sensory Attributes of Olopatadine 0.6% and Azelastine 137mcg Nasal Sprays in Patients w/Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Michael Edwards, PhD\Global Scientific Market Affairs, Alcon Research
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SMA-08-21
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Allergic Rhinitis
Keywords: rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis | interventions — Olopatadine Hydrochloride; azelastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Olopatadine 0.6% / Azelastine 137 mcg
  Interventions: Drug: Olopatadine 0.6% / Azelastine 137 mcg

INTERVENTIONS:
Drug: Olopatadine 0.6% / Azelastine 137 mcg — single dose; 2 sprays per nostril

SUMMARY:
To compare patient perceptions of the sensory attributes, including taste and aftertaste, of Olopatadine relative to azelastine when administered as a single dose in patients with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a history (at least 2 yrs) of allergic rhinitis and be symptomatic at time of enrollment
2. 18 yrs of age or older
3. Read and sign informed consent
4. Females of childbearing potential may participate if: are non-breast feeding, have negative urine pregnancy test at visit 1, agree to take urine pregnancy test upon exiting study, do not intend to become pregnant during the study, are using adequate methods of birth control.

Exclusion Criteria:

1. History of intolerance or hypersensitivity to any component of the study medications, including benzalkonium chloride.
2. Any disease or systemic disorder that may complicate or interfere with investigation or evaluation of the study medications (including but not limited to): Rhinitis medicamentosa, large obstructive nasal polyps, history (w/in last 3 months) of nasal septic ulcers, nasal surgery or nasal trauma, history or evidence of nasolacrimal drainage system malfunction, history (w/in 30 days) or evidence of sinusitis or upper or lower respiratory infection.
3. Impairment of sense of tast or smell (self reported)
4. Asthma, except for mild, intermittent asthma (nat'l Asthma guidelines)
5. Congestion, that in the opinion of the investigator, that would interfere with successful nasal drug administration/absorption
6. Patients w/a severe impairment of nasal breathing
7. Anatomic abnormalities of as identified by nasal examination
8. History of or current severe or uncontrolled cardiovascular, hepatic, renal and/or other disease/illness that could interfere w/study.
9. History of (w/in past 12 months) or ongoing clinically relevant electrolyte abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 2008- November 2008
Groups:
- Olopatadine 0.6% / Azelastine 137 Mcg: Olopatadine 0.6% / Azelastine 137 mcg
Period: Overall Study
Arm/Group | Olopatadine 0.6% / Azelastine 137 Mcg
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Olopatadine 0.6% / Azelastine 137 Mcg
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Product Preference Questionnaire for Immediate Taste
Description: Using a set of coded responses, subjects evaluated product preference in regards to immediate taste
Time Frame: 5 min post-dose
Measure: Number; unit: Percentage of participants
Arm/Group | Olopatadine 0.6% / Azelastine 137 Mcg
Number analyzed (Participants) | 102
Percentage of participants
  Preferred Azelastine Strongly | 26.47
  Preferred Azelastine Somewhat | 10.78
  Preferred Azelastine Slightly | 5.88
  Same | 15.69
  Preferred Olopatadine Slightly | 8.82
  Preferred Olopatadine Somewhat | 8.82
  Preferred Olopatadine Strongly | 23.53

2. Secondary Outcome: Taste and Aftertaste of Medication
Time Frame: 5 min, 45 min.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Olopatadine 0.6% / Azelastine 137 Mcg
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

LIMITATIONS AND CAVEATS:
Small sample size. The severity of symptoms experienced by patients may have masked their ability to detect taste and smell.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No